CLINICAL TRIAL: NCT02580604
Title: PTH And Calcium Responses to Exercise in Older Adults Experiment 2 (PACE Sr. 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 15-0878; UM1TR004399 (NIH)
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Calcium Chloride; Calcium Gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calcium Infusion followed by Saline Infusion (Experimental): All participants will have a continuous calcium infusion during exercise at their first collection visit. The second collection visit will always be a volume-matched half-normal saline infusion.
  Interventions: Drug: Calcium Chloride/Calcium Gluconate; Drug: Half-Normal Saline

INTERVENTIONS:
Drug: Calcium Chloride/Calcium Gluconate — Calcium (as either calcium chloride or calcium gluconate in half normal saline) will be delivered via IV during exercise to keep serum ionized calcium levels above baseline. The clamp is modeled after the hyperglycemic glucose clamp.
Drug: Half-Normal Saline — This is the placebo comparative infusion. Half-normal saline will be infused at the second collection visit following the identical infusion schedule determined during the calcium infusion visit.

SUMMARY:
Declines in serum calcium during exercise may cause increases in markers of bone resorption. This study will determine if preventing the decline serum ionized calcium experienced at the onset of exercise through the use of a "calcium clamp" also prevents increases in blood biomarkers associated with bone resorption.

DETAILED DESCRIPTION:
Participants will undergo two identical walking exercise sessions on a treadmill. One session will occur until continuous calcium infusion and the other will be under continuous saline infusion. C-telopeptide, parathyroid hormone, total calcium, and serum ionized calcium will be monitored to distinguish differences in bone activity under the two conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 60-80 y
* Currently taking a bisphosphonate medication

Exclusion Criteria:

* Use of medications (other than bisphosphonates) in the past 6 months known to affect bone metabolism (e.g., thiazide diuretics, oral glucocorticoids)
* Bone Mineral Density (BMD) t score < -3.0 at the total hip or lumbar spine
* Known disease or condition associated with intestinal malabsorption
* Moderate or severe renal impairment defined as an estimated glomerular filtration rate of <60 mL/min/1.73m2 based on the Modified Diet in Renal Disease (MDRD) equation
* Chronic hepatobiliary disease, defined as liver function tests (AST, ALT) >1.5 times the upper limit of normal; if such values are obtained on initial screening and thought to be transient in nature, repeated testing will be allowed
* Thyroid dysfunction, defined as an ultrasensitive TSH <0.5 or >5.0 mU/L; volunteers with abnormal TSH values will be re-considered for participation in the study after follow-up evaluation by the PCP with initiation or adjustment of thyroid hormone replacement
* Serum calcium <8.5 or >10.3 mg/dL Serum 25(OH)D <20 ng/mL; volunteers with abnormal serum 25(OH)D values may be re-considered for participation in the study if serum 25(OH)D is >20 ng/mL after vitamin D supplementation
* Uncontrolled hypertension defined as resting systolic BP >150 mmHg or diastolic BP>90 mmHg; participants who do not meet these criteria at first screening will be re-evaluated, including after follow-up evaluation by the PCP with initiation or adjustment of anti-hypertensive medications
* History of type 1 or type 2 diabetes
* Cardiovascular disease; subjective or objective indicators of ischemic heart disease (e.g., angina, ST segment depression) or serious arrhythmias at rest or during the graded exercise test (GXT) without follow-up evaluation will be cause for exclusion; follow-up evaluation must include diagnostic testing (e.g., stress echocardiogram or thallium stress test) with interpretation by a cardiologist
* Diagnosis or history of asthma

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Wherry, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Calcium Infusion First, Saline Infusion Second: Continuous calcium infusion during exercise
  Calcium Chloride/Calcium Gluconate: Calcium (as either calcium chloride or calcium gluconate in half normal saline) will be delivered via IV during exercise to keep serum ionized calcium levels above baseline. The clamp is modeled after the hyperglycemic glucose clamp.
  The second infusion will be half-normal saline following the same infusion schedule and dosing as the calcium infusion.
Period: Calcium First
Arm/Group | Calcium Infusion First, Saline Infusion Second
Started | 12
Completed | 12
Not Completed | 0
Period: Saline Second
Arm/Group | Calcium Infusion First, Saline Infusion Second
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Calcium Infusion: Continuous calcium infusion during exercise
Arm/Group | Calcium Infusion
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Parathyroid Hormone (PTH)
Description: Change in PTH will be measured from baseline to end of exercise
Time Frame: baseline, 60 minutes
Measure: Mean (95% Confidence Interval); unit: pg/mL
Groups:
- Saline Infusion: Continuous saline infusion during exercise
Arm/Group | Calcium Infusion | Saline Infusion
Number analyzed (Participants) | 12 | 12
pg/mL | 8.5 [3.5 to 13.4] | 20.0 [11.2 to 28.7]

2. Secondary Outcome: Change in C-telopeptide (CTX)
Description: Change in CTX will be measured from baseline to the end of 60 minutes of exercise
Time Frame: baseline, 60 minutes
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Calcium Infusion | Saline Infusion
Number analyzed (Participants) | 12 | 12
ng/mL | 0.01 [-0.03 to 0.06] | 0.11 [0.03 to 0.18]

3. Secondary Outcome: Change in Ionized Calcium
Description: Change in ionized calcium will be measured from baseline to the end of 60 minutes of exercise
Time Frame: baseline, 60 minutes
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Calcium Infusion | Saline Infusion
Number analyzed (Participants) | 12 | 12
mg/dL | 0.07 [0.05 to 0.20] | -0.15 [-0.29 to -0.01]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: This study was not intended to treat or prevent any disease/illness. All participants were generally healthy at time of enrollment.
Groups:
- Calcium Infusion: Continuous calcium infusion during exercise
  Calcium Chloride/Calcium Gluconate: Calcium (as either calcium chloride or calcium gluconate in half normal saline) will be delivered via IV during exercise to keep serum ionized calcium levels above baseline. The clamp is modeled after the hyperglycemic glucose clamp.
- Saline Infusion: Continuous saline infusion during exercise
  Placebo: Saline Infusion
Arm/Group | Calcium Infusion | Saline Infusion
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT02580604/Prot_SAP_000.pdf